CLINICAL TRIAL: NCT06020365
Title: Investigation of Fecal Microbiota Transplant Treatment in Chronic Intestinal Pseudo-obstruction Patients
Brief Title: Investigation of Fecal Microbiota Transplant in Chronic Intestinal Pseudo-obstruction Patients
Acronym: FMT-CIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Dean of the hospital, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT_CIPO
Record Dates: First submitted 2023-08-21; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Intestinal Pseudo-Obstruction; Fecal Microbiota Transplantation
MeSH Terms: conditions — Intestinal Pseudo-Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sequential antibiotics treatment and fecal + small intestinal microbiota transplant (Experimental)
  Interventions: Other: sequential fecal microbiota transplant combined with small intestinal fluid transplant

INTERVENTIONS:
Other: sequential fecal microbiota transplant combined with small intestinal fluid transplant — for eligible patients, the investigator use rifaximin, three times daily, 0.4 g each time, lasting 6 days followed by fecal microbiota transplant combined with small intestinal fluid transplant for 6 days. These procedures were repeated every 28 days.

SUMMARY:
Chronic Intestinal Pseudo-Obstruction (CIPO) is a rare gastrointestinal disorder that primarily affects the movement of the intestines, leading to symptoms that resemble a true bowel obstruction but without a physical blockage. This condition is characterized by impaired motility of the gastrointestinal tract, which can result in severe symptoms and complications. In previous studies, the investigator found that sequential microbiota transplantation therapy can improve clinical symptoms of chronic pseudo-obstruction. Building on this foundation, the current study further investigates the effects of sequential interventions involving intestinal cleansing, small intestine bacterial treatment, fecal microbiota transplantation, and nutritional therapy on the short-term and long-term clinical symptom improvement in patients. Additionally, the investigator aim to elucidate the changes in gut microbiota phenotypes before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. aged over 18 years old;
2. met the current diagnosis criteria for Chronic Intestinal Pseudo-obstruction;
3. can tolerate nasojejunal tube and complete full course of FMT treatment;
4. the clinical data are relatively complete and there is follow-up available for evaluation

Exclusion Criteria:

1. accompanied by chronic wasting diseases such as malignant tumor and hyperthyroidism;
2. associated with gastrointestinal organic diseases such as short bowel syndrome, intestinal fistula, and inflammatory bowel disease; c) severe destruction of the intestinal mucosa, severe immunosuppression, combined with severe systemic infection; d) Intervention with antibiotics during treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Enteral Nutrition Tolerance | 8 weeks
  the maximal amount of enteral nutrition allowed daily

SECONDARY OUTCOMES:
Nutrition Status | 52 weeks
  intersectional muscle and fat area measurements by quantitative computed tomography

OTHER OUTCOMES:
Need for surgery | 52 weeks
  Surgical interventions are performed due to intestinal nutritional intolerance, including procedures such as nutritional ostomy, decompression ostomy, and intestinal resection.
Changes of both colerectal and small intestinal microbiota profile | 8 weeks
  Both colorectal and small intestinal bacteria profile before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes